CLINICAL TRIAL: NCT02225041
Title: Sedation Strategy and Cognitive Outcome After Critical Illness in Early Childhood
Acronym: RESTORE-cog
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01HD074757-01A1 (NIH); 1R01HD074757-01A1 (NIH)
Record Dates: First submitted 2014-07-25; First posted 2014-08-25 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Intellectual Disability; Perceptual Disorders; Memory Disorders
Keywords: intensive care; critical care; child; family; survivors
MeSH Terms: conditions — Intellectual Disability; Perceptual Disorders; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the relationships between sedative exposure during pediatric critical illness and long-term neurocognitive outcomes. We will test for drug- and dose-dependent relationships between sedative exposure and neurocognitive outcomes along the early developmental spectrum and will control for baseline and environmental factors, as well as the severity and course of illness.

Hypotheses:

1. Greater exposure to benzodiazepines and/or ketamine will be associated with lower IQ even when controlling for severity of illness, hospital course, and baseline factors. In addition, benzodiazepines and/or ketamine will negatively affect other aspects of neurocognitive function.
2. Younger children exposed to benzodiazepines and/or ketamine will have worse neurocognitive outcomes than older children with similar sedative exposure and severity of illness.

DETAILED DESCRIPTION:
Ensuring the safety and comfort of the more than 100,000 critically ill infants and young children supported on mechanical ventilation in the US each year is integral to the practice of pediatric critical care. Humane care of these young patients requires the use of sedating medications, most commonly combinations of opioids and benzodiazepines. Unfortunately, sedative use also carries risk. Animal studies found that even transient administration of benzodiazepines and other sedatives during periods of developmental synaptogenesis caused widespread neuronal apoptosis and residual learning and memory deficits. Sedation is administered for days to weeks in >90% of acutely-ill, ventilated infants and children. Thus, a commonly used treatment in critically ill young children may itself have detrimental, age-dependent long-term effects.

An opportunity to increase the understanding of the long-term cognitive effects of sedation during critical illness in children has been provided by the cluster randomized, controlled trial of a sedation protocol, Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE), U01 HL086622, PI Curley, 31 sites, n=2,816. This trial determined whether the trial's sedation protocol used at intervention sites decreased the duration of mechanical ventilation and sedative exposure among children with acute respiratory failure due to a primary pulmonary process. Control sites continued usual sedation practice. We collected detailed data on doses and durations of sedative medications, in-hospital course, and post-discharge quality of life.

The purpose of RESTORE-cognition is to determine the relationships between sedative exposure during pediatric critical illness and long-term neurocognitive outcomes. We will assess multiple domains of neurocognitive function 2.5-5 years post-discharge in 500 RESTORE subjects with normal baseline cognitive function aged 2 weeks to 8 years at pediatric intensive care unit admission. In addition, we will study 310 matched, healthy siblings of RESTORE subjects to provide data on an unexposed group with similar baseline biological characteristics and environment. Our goal is to increase our understanding of the relationships between sedative exposure, critical illness, and long-term neurocognitive outcomes in infants and young children.

ELIGIBILITY:
Inclusion Criteria:

RESTORE subjects

* Age ≤8 years and PCPC=1 at RESTORE PICU admission
* PCPC ≤3 at RESTORE hospital discharge Sibling control subjects

Inclusion criteria:

* Age 4 to 17 years at time of testing
* PCPC=1
* Same biological parents as primary subject
* Lives with the primary subject

Exclusion Criteria:

RESTORE subjects

* Hospital readmission that includes MV and sedation
* History of cardiac arrest, traumatic brain injury (TBI) with loss of consciousness, genetic disorder, premature birth <32 weeks gestational age, or birth weight <2500 g Sibling control subjects
* Adopted or step siblings
* History of MV and sedation, receipt of general anesthesia, cardiac arrest, TBI with loss of consciousness, genetic disorder, premature birth <32 weeks gestational age, or birth weight <2500 gm.

Ages: 30 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: RESTORE subjects who consented for 6-month follow-up with normal baseline cognitive function aged 2 weeks to 8 years at PICU admission. In addition, we will study matched, healthy siblings of these subjects to provide data on an unexposed group with similar baseline biological characteristics and environment. If more than one sibling meets enrollment criteria, the one closest in age will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function at 2.5 years post-ICU discharge, as assessed using standardized tests of attention, processing speed, learning and memory, visual-spatial skills, motor skills, language, executive function, IQ, and behavior | 2.5 to 5 years post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, RN, PhD, Principal Investigator — University of Pennsylvania; R. Scott Watson, MD, Principal Investigator — Seattle Childrens Hospital
Locations (31):
- United States (31):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University Medical Center, The University of Arizona, Tucson, Arizona
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital at University of California San Francisco Medical Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Holtz Children's Hospital, Miami, Florida
  - Florida Hospital for Children, Orlando, Florida
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - University of Maryland Hospital for Children, Baltimore, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - University of Massachusetts Memorial Children's Medical Center, Worcester, Massachusetts
  - C. S. Mott Children's Hospital of the University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Medical City Children's Hospital, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Curley MAQ, Watson RS, Cassidy AM, Burns C, Delinger RL, Angus DC, Asaro LA, Wypij D, Beers SR; RESTORE-cognition Study Investigators. Design and rationale of the "Sedation strategy and cognitive outcome after critical illness in early childhood" study. Contemp Clin Trials. 2018 Sep;72:8-15. doi: 10.1016/j.cct.2018.07.004. Epub 2018 Jul 11. PMID 30017814